CLINICAL TRIAL: NCT06816056
Title: Safety and Efficacy of Manual Therapy in the Treatment of Haemophilic Arthropathy of the Ankle. A Randomised Multicentre Clinical Trial
Brief Title: Manual Therapy in Hemophilic Arthropathy of the Ankle
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Principal Investigator, Rubén Cuesta-Barriuso, Principal Investigator, Investigación en Hemofilia y Fisioterapia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HE-ANKLEran
Record Dates: First submitted 2025-02-03; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Hemophilia A
Keywords: Hemophilic arthropathy; Ankle; Manual therapy; Joint pain
MeSH Terms: conditions — Hemophilia A; Arthralgia | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The intervention will last 3 weeks, with a periodicity of 1 weekly sessions. In total there will be 3 sessions lasting 50 minutes.
  The techniques will be: global passive mobilisation, calcaneocuboid mobilisation, talus-navicular mobilisation, talar manipulation, tibial displacement manipulation, tibiotarsal decompression, plantar fascia induction, tibiotarsal unwinding traction technique and triceps surae induction technique
  Interventions: Other: Manual Therapy
- Control group (Placebo Comparator): The patients included in the control group will receive the same physiotherapy intervention in the form of a placebo. The physiotherapist in charge of this intervention will perform the same number of techniques but without applying sliding stimuli, myofascial induction or manipulation. The hands will be positioned in the same way and the times per technique will be the same as in the techniques of the experimental group.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Manual Therapy — The patients included in the experimental group will receive a 50-minute physiotherapy intervention involving global passive mobilisation, calcaneocuboid mobilisation, talus-navicular mobilisation, talar manipulation, tibial displacement manipulation, tibiotarsal decompression, plantar fascia induction, tibiotarsal unwinding and triceps surae induction techniques
  Arms: Experimental group
Other: Placebo — The patients included in the control group will receive a 50-minute physiotherapy intervention in which the physiotherapist's hands and the times per technique will be the same as in the experimental group, but without applying any sliding, mobilisation or manipulation
  Arms: Control group

SUMMARY:
Introduction: Haemophilic ankle arthropathy manifests as functional (deficit in muscle strength, mobility and proprioception), intra-articular degenerative alterations and chronic pain. Manual therapy techniques are characterised by treating the soft tissues with the aim of modifying their density, relieving pain, reducing tissue sensitivity and improving the ranges of mobility. The objective is to evaluate the safety and effectiveness of a manual therapy protocol in patients with haemophilic ankle arthropathy.

Methods: Randomised crossover clinical trial. 13 patients with haemophilic ankle arthropathy from different regions of Spain will be recruited and randomised into two study groups (experimental and control). Each session of the experimental group will last 50 minutes, with 1 physiotherapy session per week for a period of 3 weeks. Patients will be evaluated at the beginning of the study, after the intervention and after a follow-up period of 4 weeks. The treatment programme includes 10 techniques that must be administered bilaterally. The study variables are the frequency of ankle haemarthrosis, range of movement, pressure pain threshold, pain intensity, joint status, biomechanical analysis of gait and balance, functionality and kinesiophobia.

Expected results: To evaluate the safety of manual therapy in patients with haemophilia. To observe changes in pain, mobility, joint condition, stability and functionality of the ankle, and kinesiophobia.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with haemophilia A and B
* With severe haemophilia phenotype (<1% FVIII/FIX)
* Over 18 years of age
* With a medical diagnosis of ankle arthropathy and with clinical assessment using the Hemophilia Joint Health Score
* On prophylactic or on-demand treatment with coagulation factor VIII/FIX concentrates

Exclusion Criteria:

* Patients with neurological or cognitive disorders that prevent them from understanding the questionnaires and physical tests
* Failure to sign the informed consent document

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2025-02-05 (Estimated); Primary Completion 2025-07-21 (Estimated); Study Completion 2025-07-25 (Estimated)

PRIMARY OUTCOMES:
Change from baseline hemarthrosis after treatment and at four weeks | Screening visit, within the first seven days after treatment and after four weeks follow-up visit
  A self-registration will be used to evaluate the frequency of bleeding, and thus the safety of the technique. This self-registration will be given to each patient at the beginning of the study and they must fill in the number of hemarthrosis and their main characteristics: date, origin (traumatic or spontaneous). The self-registration will be delivered to the evaluator in each of the study evaluations (post-treatment and follow-up).

SECONDARY OUTCOMES:
Change from baseline pressure pain threshold after treatment and at four weeks | Screening visit, within the first seven days after treatment and after four weeks follow-up visit
  Using a pressure algometer (model Wagner FPN100) we will measure the pain threshold to pressure, at the level of the joint and at a distance (in another part of the body). This device measures in Newton/cm2 the pressure at which the subject perceives pain under pressure. Pressure will be applied to the chosen point, which will be increased at a rate of approximately 50 kPa/s until the patient informs us that the sensation is starting to become painful. The lateral and medial malleoli of the ankle will be evaluated
Change from baseline joint status after treatment and at four weeks | Screening visit, within the first seven days after treatment and after four weeks follow-up visit
  Change from knee and ankle joint status during treatment and follow-up period at four weeks. Measurement instrument: Haemophilia Joint Health Score (scale 0-20).
Change from baseline range of motion after treatment and at four weeks | Screening visit, within the first seven days after treatment and after four weeks follow-up visit
  Change from range of movement of ankle during treatment and follow-up period at four weeks. The range of motion of the ankle joint will be measured using a universal goniometer, using the protocol for measuring joint motion described by the American Academy of Orthopaedic Surgeons
Change from baseline joint pain after treatment and at four weeks | Screening visit, within the first seven days after treatment and after four weeks follow-up visit
  Change in ankle intensity during treatment and the four-week follow-up period. Ankle joint pain intensity will be measured using the visual analogue scale with a range of 0 to 10 points, where the higher the score, the greater the perception of joint pain
Change from baseline functional capacity after treatment and at four weeks | Screening visit, within the first seven days after treatment and after four weeks follow-up visit
  Change in functional capacity during treatment and the four-week follow-up period. Functional capacity will be measured using the 2-Minutes Walking Test. The maximum distance that patients can cover in a period of six minutes walking as fast as possible will be measured. The unit of measurement is the metre, where the greater the distance, the better the functional capacity.
Change from baseline kinesiophobia after treatment and at four weeks | Screening visit, within the first seven days after treatment and after four weeks follow-up visit
  Change in kinesiophobia during treatment and the four-week follow-up period. Fear of movement will be measured using the Tampa scale, which consists of 11 items on a 4-point Likert scale, with responses ranging from 1 (strongly disagree) to 4 (strongly agree). The lowest possible score, 11, denotes insignificant or non-existent kinesiophobia. The highest possible score, 44, denotes a severe fear of feeling pain when moving

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Universidad de Oviedo
Locations (1):
- Universidad Católica San Antonio, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No